CLINICAL TRIAL: NCT04072081
Title: Multicenter, Randomized, Open and Controlled Study of Drug-coated Balloon Versus Drug-eluting Stent in the Treatment of Coronary Artery Lesions in STEMI Patients in De Novo Coronary Lesions
Brief Title: Drug-coated Balloon Versus Drug-eluting Stent in the Treatment of Coronary Artery Lesions in STEMI Patients in De Novo Coronary Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital,School of Medicine,Zhejiang University &Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT014
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated ballon (Experimental): Treatment of in suit coronary lesions with drug-coated balloon
  Interventions: Device: Drug-coated balloon
- Drug-eluting stent (Active Comparator): Treatment of in suit coronary lesions with drug-eluting stent
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-coated balloon — Treatment of in suit coronary lesions with drug-coated balloon
  Arms: Drug-coated ballon
Device: Drug-eluting stent — Treatment of in suit coronary lesions with drug-eluting balloon
  Arms: Drug-eluting stent

SUMMARY:
The study aims to find a DCB treatment for STEMI patients can achieve early and mid-term functional outcomes that are not inferior to DES, and realize the strategy of intervention without implantation.

DETAILED DESCRIPTION:
The main objective of this study is to compare a Drug-coated Ballon with Drug-eluting stent in the treatment of coronary arty lesions in STEMI patients in de novo coronary lesions.The study aims to find a DCB treatment for STEMI patients can achieve early and mid-term functional outcomes that are not inferior to DES, and realize the strategy of intervention without implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical criteria 1)over 18 years old 2)Angiographic confirmation of acute myocardial infarction 3)EKG prompts STEM basis 4)Sign informed consent
2. Angiographic criteria 1)In situ coronary artery disease 2)The reference diameter of the target vessel was 2.5-3.5 mm and the length was less than 28 mm 3)Visual examination showed that the diameter of lesions in criminals was narrower than or equal to 80%.

Exclusion Criteria:

1.Clinical criteria

1. LVEF<30%
2. Killip grading is greater than 3
3. Significant abnormalities in hemorrhagic quality or known coagulation function
4. History of intracranial tumors, aneurysms, arteriovenous malformations or cerebral hemorrhage;There was a history of stroke or TIA in 6 months and gastrointestinal bleeding in 2 months.Major operations were performed within 6 weeks.Recent or known platelets < 100,000/mm3 or hemoglobin < 10 g/dL.
5. Planned elective surgery may lead to early discontinuation of ADP receptor antagonists
6. The expected survival time of patients with other systemic diseases, such as malignant tumors is less than 1 year 2.Angiographic criteria

1)Left main lesion 2)The grade of dissection is greater than or equal to grade C lesions. 3)Coronary artery bridge lesions 4)In-stent restenosis 5)Severe stenosis of non-criminal lesions requiring selective treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Late luminal loss (LLL) | 9 months
  LLL was the difference between the in-segment minimal lumen diameter after the procedure and at angiographic follow-up, as evaluated by quantitative coronary angiography

SECONDARY OUTCOMES:
Restenosis rate (RR) | 12-24 months
  in-stent restenosis
Target lesion failure (TLF) | 12-24 months
  The occurrence of cardiac death, target vessel myocardial infraction and target vessel revascularization
Target lesion thrombosis | 12-24 months
  Thrombus was classified as definite, probable, or possible, according to the definitions provided by the Academic Research Consortium (ARC). Regarding timing, ST was defined as early (<30 days), late (30 days to 1 year), or too late (>1 year)
MACE | 12-24 months
  Non-fatal acute myocardial infarction, severe arrhythmia, heart failure, cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Jun, PhD, Study Director — Second Affiliated Hospital Zhejiang University School of Medicine